CLINICAL TRIAL: NCT02294799
Title: Magnetic Ressonance Imaging Evaluation of Articular Disc Position in TMD Subjects After Mandibular Mobilization. A Double Blind, Randomized, Placebo-controlled Study
Brief Title: Magnetic Ressonance Imaging of Temporomandibular Joint
Acronym: MRITMJ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Ap. Biasotto-Gonzalez (Other)
Responsible Party: Sponsor-Investigator, Daniela Ap. Biasotto-Gonzalez, Phd, University of Nove de Julho
Organization: University of Nove de Julho (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YEH1984
Record Dates: First submitted 2013-04-09; First posted 2014-11-19 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Temporomandibular Joint Dysfunction
Keywords: Temporomandibular Joint Disorders; Magnetic Ressonance Imaging; Complementary Therapy; Physical Therapy Modalities.
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Other): TMD diagnosed sujects that will receive the mobilization treatment
  Interventions: Other: Intervention Group
- Placebo Group (Placebo Comparator): TMD diagnosed sujects that will receive the placebo treatment
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: Intervention Group — Grade 1, Nonspecific Mandibular Mobilization
  Other Names: Mandibular Mobilization
  Arms: Intervention Group
Other: Placebo group — Nonspecific Mandibular Movement.
  Other Names: Placebo Mandibular Mobilization
  Arms: Placebo Group

SUMMARY:
Background: Among the instrumental devices that have been proposed over the years to integrate the clinical evaluation of temporomandibular joint disorders (TMD), imaging techniques are the most studied, showing that magnetic resonance imaging (MRI) is the technique most need to describe the anatomy of the TMJ and to evaluate the correlation of imaging findings with the clinical diagnosis . Despite the amount available studies on the use of MRI for evaluation of TMJ disorders and treatments, there is a lack of studies that evaluate the imaging findings after physical therapy. Purpose: To evaluate the influence of nonspecific mandibular mobilization about the positioning of the articular disc by MRI in individuals with TMD diagnosis of anterior disc displacement with and without reduction according to the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD). Analyze the behavior of pain through the numerical scale of pain assessment (END) at baseline and after each treatment session, the quality of life of individuals with TMD at baseline, immediately, three and six months after the treatment sessions by the World Health Organization Quality of Life Assessment (WHOQOL - BREF), and The Patient's Specific Functional Scale (PSFS) at baseline and after treatment. The treatment will be performed three times a week during four weeks. Metodology: This is a randomized, placebo controlled, blind study designed to assess the effects of techniques nonspecific mandibular mobilization x placebo. Individuals will be randomized and divided into two groups: Group A (intervention) and Group B (placebo). Statistic analysis: The positioning of the articular disc, extracted through the use of MRI, will be considered the primary outcome and, as a secondary outcome will be assessed the quality of life, pain and function after treatment. The adherence of the data to a Gaussian curve will be verified by the Shapiro-Wilk and the data are expressed as mean values and standard deviation. Two-way repeated measures analysis of variance with Bonferroni post hoc test will be used for inter-and intra-group comparisons. The significance level is adjusted p ≤ 0.05.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind study designed to verify the effects of nonspecific mandibular mobilization techniques x placebo

ELIGIBILITY:
Inclusion Criteria:

* TMD diagnosed subjects by RDC / TMD confirmed by the MRI findings,
* with anterior disk displacement with or without reduction,
* with full dentition (excluding third molars).

Exclusion Criteria:

* Subjects diagnosed TMD exclusively muscular;
* with posterior and / or medial displacement of the disc;
* showing systemic diseases that affect the joints and / or masticatory muscles;
* neuromuscular diseases;
* hypo / condylar hyperplasia;
* making use of any type of dental prosthesis;
* are in orthodontic and / or physical therapy;
* showing neurological or behavioral disorders that preclude the achievement of MRI and/or
* a history of previous TMJ surgery.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Articular Disc Positioning (Measured by the Magnetic Ressonance Imaging) | Baseline (day 1) and after 4 weeks of treatment performed 3 times a week.
  Measured by the Magnetic Ressonance Imaging

SECONDARY OUTCOMES:
Clinical Symptoms (Measured by END) | Baseline (day 1) and after 4 weeks of treatment performed 3 times a week.
  Measured by numerical scale of pain assessment (END)
Functionality (Mesuread by "The Patient´s Specific Funcional Scale - HORN, 2012) | Baseline (day 1) and after 4 weeks of treatment performed 3 times a week.
  Mesuread by "The Patient´s Specific Funcional Scale - HORN, 2012
Quality of life (Whoqol-bref) | Baseline (day 1) and after 4 weeks of treatment (performed 3 times a week), 3 and 6 months follow up
  Whoqol-bref

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ap Biasotto-Gonzalez, PHD, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Ahmad M, Hollender L, Anderson Q, Kartha K, Ohrbach R, Truelove EL, John MT, Schiffman EL. Research diagnostic criteria for temporomandibular disorders (RDC/TMD): development of image analysis criteria and examiner reliability for image analysis. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Jun;107(6):844-60. doi: 10.1016/j.tripleo.2009.02.023. PMID 19464658
- [Background] de Lucena LB, Kosminsky M, da Costa LJ, de Goes PS. Validation of the Portuguese version of the RDC/TMD Axis II questionnaire. Braz Oral Res. 2006 Oct-Dec;20(4):312-7. doi: 10.1590/s1806-83242006000400006. PMID 17242791
- [Background] Gray RJ, Quayle AA, Hall CA, Schofield MA. Physiotherapy in the treatment of temporomandibular joint disorders: a comparative study of four treatment methods. Br Dent J. 1994 Apr 9;176(7):257-61. doi: 10.1038/sj.bdj.4808429. PMID 8186034
- [Background] Furto ES, Cleland JA, Whitman JM, Olson KA. Manual physical therapy interventions and exercise for patients with temporomandibular disorders. Cranio. 2006 Oct;24(4):283-91. doi: 10.1179/crn.2006.044. PMID 17086858
- [Background] Ohnuki T, Fukuda M, Nakata A, Nagai H, Takahashi T, Sasano T, Miyamoto Y. Evaluation of the position, mobility, and morphology of the disc by MRI before and after four different treatments for temporomandibular joint disorders. Dentomaxillofac Radiol. 2006 Mar;35(2):103-9. doi: 10.1259/dmfr/25020275. PMID 16549437
- [Background] Horn KK, Jennings S, Richardson G, Vliet DV, Hefford C, Abbott JH. The patient-specific functional scale: psychometrics, clinimetrics, and application as a clinical outcome measure. J Orthop Sports Phys Ther. 2012 Jan;42(1):30-42. doi: 10.2519/jospt.2012.3727. Epub 2011 Oct 25. PMID 22031594
- [Background] Aigner M, Forster-Streffleur S, Prause W, Freidl M, Weiss M, Bach M. What does the WHOQOL-Bref measure? Measurement overlap between quality of life and depressive symptomatology in chronic somatoform pain disorder. Soc Psychiatry Psychiatr Epidemiol. 2006 Jan;41(1):81-6. doi: 10.1007/s00127-005-0997-8. Epub 2006 Jan 1. PMID 16341612
- [Background] El Hage Y, Politti F, de Sousa DF, Herpich CM, Gloria IP, Gomes CA, Amaral AP, de Melo NC, da Silva TC, Arruda EE, Amorim CF, Gadotti IC, Gonzalez TO, Berzin F, Bussadori SK, Garcia MB, Barbosa BR, Biasotto-Gonzalez DA. Effect of mandibular mobilization on electromyographic signals in muscles of mastication and static balance in individuals with temporomandibular disorder: study protocol for a randomized controlled trial. Trials. 2013 Oct 1;14:316. doi: 10.1186/1745-6215-14-316. PMID 24083628
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Emshoff R, Brandlmaier I, Gerhard S, Strobl H, Bertram S, Rudisch A. Magnetic resonance imaging predictors of temporomandibular joint pain. J Am Dent Assoc. 2003 Jun;134(6):705-14. doi: 10.14219/jada.archive.2003.0256. PMID 12839406
- [Background] Emara AS, Faramawey MI, Hassaan MA, Hakam MM. Botulinum toxin injection for management of temporomandibular joint clicking. Int J Oral Maxillofac Surg. 2013 Jun;42(6):759-64. doi: 10.1016/j.ijom.2013.02.009. Epub 2013 Mar 26. PMID 23538215